CLINICAL TRIAL: NCT01821911
Title: Phase 4 Study of Speeda® Rabies Vaccine for Human Use
Brief Title: The Post-Marketing Safety and Immunogenicity Research of Speeda® Rabies Vaccine for Human Use
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BJCDPC-5
Record Dates: First submitted 2013-03-27; First posted 2013-04-01 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2013-04

CONDITIONS: Rabies Vaccine Allergy; Vaccination Adverse Event; Anti-D Antibodies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zagreb2-1-1 (Experimental): Injection on day 0、7、21
  Interventions: Biological: Zagreb2-1-1; Biological: Essen
- Essen (Active Comparator): Injection on day 0、3、7、14、28
  Interventions: Biological: Zagreb2-1-1; Biological: Essen

INTERVENTIONS:
Biological: Zagreb2-1-1 — Injection on day 0、7、21
Biological: Essen — Injection on day 0、3、7、14、28

SUMMARY:
The objective of this study was to achieve the post-marketing safety and immunogenicity research of Speeda® rabies vaccine for human use from Chengda Bio

DETAILED DESCRIPTION:
The aim of the research is to compare the two immune procedures. The investigators plan to enroll 10500 participants signed the informed consent who separately inject by Zagreb or Essen procedure.

ELIGIBILITY:
Inclusion Criteria:

* Parent/legal acceptable representatives of children or the adult participants are willing and able to understand the protocol requirements and provide informed consent signed
* Participant is considered to be in good health including the body and mental status on the basis of reported medical history and limited physical examination and live in local ≥ 12 months
* Participant body temperature ≤ 37.0℃
* Participant without preventive inoculation of rabies vaccine(only limited in immunogenicity subgroup)

Exclusion Criteria:

* Three-level exposure
* Known allergy to any constituent of the vaccine
* Reported the history of allergies, convulsions, epilepsy, mental illness and brain disease and clear serious systemic reaction
* Known bleeding disorder or suspected impairment of immunologic function, or receipt of immunosuppressive therapy or immunoglobulin since birth
* Participation in any other interventional clinical trial
* An acute illness with or without fever (temperature > 37.0℃) in the latest week preceding enrollment in the trial
* Inoculated other vaccines, immunoglobulin or investigational drugs within 4 weeks prior to participation in the study
* Reported clearly the infection of the upper respiratory tract with 6 months Clinical Manifestation of Metabolic, blood system, lungs, heart, the gastrointestinal tract, nervous system, kidneys, urinary system, endocrine, liver disease or malignant tumor
* Any condition which, in the opinion of the investigator, would pose a health risk to the subject or interfere with the vaccine

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10500 (Actual)
Dates: Start 2012-07; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Incidence Rate of Adverse Events of the rabies vaccine each injection | 2 years

SECONDARY OUTCOMES:
Antibody titre of the subject on 0、7、14、42、180、365 | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Nianmin Shi, Principal Investigator — Beijing Chaoyang District Centers for Disease Control and Prevention
Locations (3):
- China (3):
  - Guangdong Centers for Disease Control and Prevention, Zhaoqing, Guangdong
  - Wuhan Centers for Disease Control and Prevention, Wuhan, Hubei
  - Beijing Chaoyang District Centers for Disease Control and Prevention, Beijing

REFERENCES:
- [Derived] Li L, Xu J, Zhang J, Wang F, Cai J, Yang L, Zhu Z, Bai Y, Jia B, Ma J, Shi N, Li S. Immunogenicity and immune persistence of Zagreb 2-1-1 regimen of rabies vaccine in Chinese healthy individuals: A randomized, parallel-controlled of homologous vaccine with different immune procedure study. Hum Vaccin Immunother. 2024 Dec 31;20(1):2403177. doi: 10.1080/21645515.2024.2403177. Epub 2024 Oct 2. PMID 39358206
- [Derived] Shi N, Zhang Y, Zheng H, Zhu Z, Wang D, Li S, Li Y, Yang L, Zhang J, Bai Y, Lu Q, Zhang Z, Luo F, Yu C, Li L. Immunogenicity, safety and antibody persistence of a purified vero cell cultured rabies vaccine (Speeda) administered by the Zagreb regimen or Essen regimen in post-exposure subjects. Hum Vaccin Immunother. 2017 Jun 3;13(6):1-8. doi: 10.1080/21645515.2017.1279770. Epub 2017 Jan 25. PMID 28121231